CLINICAL TRIAL: NCT00371462
Title: PDA+: A Personal Digital Assistant for Obesity Treatment
Acronym: PDA+
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: PI no longer has an appointment and has seperated from Hines VAH and project was not transferred to another PI?
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: F4429-I
Record Dates: First submitted 2006-08-31; First posted 2006-09-04 (Estimated); Results first posted 2016-10-07 (Estimated); Last update posted 2016-10-07 (Estimated); Status verified 2016-08

CONDITIONS: Obesity; Pain
Keywords: intervention study; technology; weight loss
MeSH Terms: conditions — Obesity; Pain; Weight Loss

ARMS (2):
- Arm 1 (Active Comparator): MOVE! level 2 group weight loss counseling, the VA standard of care alone (Standard Care);
  Interventions: Behavioral: Use of PDA + support to reduce weight and pain
- Arm 2 (Experimental): MOVE! level 2 + Personal Digital Assistant decision support tool (PDA) (Treatment)
  Interventions: Behavioral: MOVE! level 2 group weight loss counseling

INTERVENTIONS:
Behavioral: Use of PDA + support to reduce weight and pain — participants will attend the MOVE! group, record their food, activity, mood, pain, and weight daily via a PDA. Participants will be assigned a coach to help them set physical activity and calorie goals in order to produce a weight loss of .5%-1% per week on average over the course of 6 months. Participants will continue to log using the PDA during the 2nd 6-months for follow-up. They will also be asked to attend assessments at 3, 6, 9, and 12 months.
  Arms: Arm 1
Behavioral: MOVE! level 2 group weight loss counseling — Participants will attend the MOVE! group and will be asked to complete assessments at 3, 6, 9, and 12 months.
  Arms: Arm 2

SUMMARY:
The purpose of this study is to determine whether including a PDA decision support tool plus distance support enhances the outcomes attainable by the MOVE2! (Managing Obesity for Veterans Everywhere) standard care alone. Primary hypotheses are that obese patients with chronic pain who are randomized to MOVE2! + PDA + Support will a) lose more weight by 6 months, b) show greater maintenance of weight loss at 12 months, and c) display greater reduction in pain intensity and pain-related disability than those randomized to Standard Care. Secondary hypotheses are that MOVE2! + PDA + Support, compared to Standard Care will result in: a) improved quality of life, b) greater treatment adherence, and c) reduced care utilization.

DETAILED DESCRIPTION:
An obesity epidemic is gaining momentum in the U.S. and the VA in particular. Among Veterans receiving care at VA outpatient centers in the year 2000, the prevalence of overweight was 73% and obesity was 33%. Obesity is an expensive condition partly because it contributes to the development of other chronic diseases. In addition to its adverse medical consequences, obesity takes a toll on quality of life. In general and among veterans specifically, obesity is associated with chronic pain conditions. Pain and obesity in combination adversely affect health-related quality of life and increase care utilization. To treat obesity, VA patient services has implemented MOVE! (Managing Obesity for Veterans Everywhere), a nationwide, pre-inpatient, pre-surgical standard of care. MOVE! Level 2 (MOVE2!), the platform for this study, enrolls in group treatment patients who are ready to make behavioral changes in diet and physical activity. The current study interfaces with and adds to MOVE2! treatment in order to maximize utility and sustainability in VA. The intervention in the current study involves provision of a personal digital assistant (PDA), a hand-held computer decision support tool to self-regulate diet and activity along with staff support (via telephone or e-mail per patient's preference).

Experimental Design. The current study is a 2-group prospective randomized controlled trial comparing the effects of (1) Standard Care: MOVE2! group weight loss counseling alone and (2) MOVE2! + PDA + Support. Specific aims are to enroll from VA primary care a sample of 150 obese patients who meet study criteria for chronic pain and are ready to make behavioral changes, including enrolling in MOVE2!. Primary outcomes (weight and pain) and secondary outcomes (quality of life, treatment adherence, healthcare utilization) will be measured every 3 months (baseline, treatment months 3 and 6, and follow-up months 9 and 12). Before beginning the current study, we will conduct two types of formative research. Part 1A: We will recruit 15 Veterans who are obese and have chronic pain for the purpose of pilot testing the PDA. Veterans will participate in one focus group before and one after they use the PDA for one week. Part 1B: We will also conduct focus groups with 10 MOVE! personnel and 10 staff who work in Hines Primary Care Clinic to identify perceived needs and barriers regarding implementing our PDA intervention.

Objective & Hypotheses. To determine whether the provision of a PDA decision support tool plus distance support enhance the outcomes attainable by the MOVE2! standard care alone. Primary hypotheses are that obese patients with chronic pain who are randomized to MOVE2! + PDA + Support will a) lose more weight by 6 months, b) show greater maintenance of weight loss at 12 months, and c) display greater reduction in pain intensity and pain-related disability than those randomized to Standard Care. Secondary hypotheses are that MOVE2! + PDA + Support, compared to Standard Care will result in: a) improved quality of life, b) greater treatment adherence, and c) reduced care utilization.

Data Analysis. Outcomes will be analyzed longitudinally on an intent to treat basis. The general analytic approach will be to use longitudinal mixed-effects regression models implemented via SAS PROC MIXED. Stratification variables (age, BMI, gender) will be included in all analyses.

ELIGIBILITY:
Inclusion Criteria:

* Patients with BMI >25 will be recruited from the primary care clinics at Hines Hospital VAMC. Enrollment of patients with this BMI criteria allows comparability with other obesity behavioral treatment trials. The enrollment policy is also consistent with the 2005 VA/DoD Practice Guideline that recommends obesity treatment for all Veterans with BMI >25.
* Male or female Veterans
* Age >18
* With chronic pain (Numeric Rating Scale of pain intensity [NRS-I] > 4 for > 6 months prior to enrollment)
* Ready to make a weight loss effort involving diet and activity change
* Able to communicate comfortably in English.
* The primary pain complaint must be possibly related to obesity (e.g., back, knee, leg, neck, arm, or full-body pain, and not exclusively headache or cancer-related pain).

Exclusion Criteria:

* Has an active eating disorder or substance abuse disorder --Participating in another VA-funded research project -Significant cognitive or sensorimotor impairment precluding use of the PDA
* Already participating in a structured diet or exercise program or plans to begin such a program outside the study during the next year; requires use of an assistive device for mobility
* At risk for adverse cardiovascular events with moderate intensity activity
* Plans to relocate within the upcoming year

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2007-10; Primary Completion 2009-09 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Edward Hines, Jr. VA Hospital, Hines, Illinois, United States

REFERENCES:
- [Derived] Spring B, Duncan JM, Janke EA, Kozak AT, McFadden HG, DeMott A, Pictor A, Epstein LH, Siddique J, Pellegrini CA, Buscemi J, Hedeker D. Integrating technology into standard weight loss treatment: a randomized controlled trial. JAMA Intern Med. 2013 Jan 28;173(2):105-11. doi: 10.1001/jamainternmed.2013.1221. PMID 23229890
- [Derived] Duncan JM, Janke EA, Kozak AT, Roehrig M, Russell SW, McFadden HG, Demott A, Pictor A, Hedeker D, Spring B. PDA+: A Personal Digital Assistant for Obesity Treatment - an RCT testing the use of technology to enhance weight loss treatment for veterans. BMC Public Health. 2011 Apr 11;11:223. doi: 10.1186/1471-2458-11-223. PMID 21481253

RESULTS

PARTICIPANT FLOW:
Groups:
- + Mobile: Participants were provided standard-of-care (participation in VA MOVE program) plus a connective mobile technology system. Participants were provided a personal digital assistant to self-monitor diet and physical activity; they also received biweekly coaching calls for 6 months.
- Standard-of-care: Participants were provided standard-of-care (participation in VA MOVE program) for weight loss.
Period: Overall Study
Arm/Group | + Mobile | Standard-of-care
Started | 35 | 35
Completed | 27 | 27
Not Completed | 8 | 8
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Other | 7 | 8

BASELINE CHARACTERISTICS:
Population: One subject withdrew from the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1 | Arm 2 | Total
Number analyzed (Participants) | 34 | 35 | 69
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.7 (13.5) | 57.7 (10.2) | 57.7 (11.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 10
  Male | 29 | 30 | 59
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 3 | 4
  Not Hispanic or Latino | 33 | 32 | 65
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 9 | 8 | 17
  White | 25 | 27 | 52
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 34 | 35 | 69
Weight (kg) [Mean (Standard Deviation); unit: kg] | 113.7 (16.1) | 110.1 (15.1) | 111.1 (15.6)
BMI [Mean (Standard Deviation); unit: kg/m2] | 36.9 (5.4) | 35.8 (3.8) | 36.3 (4.6)
Waist circumference (cm) [Mean (Standard Deviation); unit: cm] | 120.4 (14.0) | 120.4 (8.9) | 120.4 (11.7)

OUTCOME MEASURES:

1. Primary Outcome: Weight (Measured at Assessment Visits) and Pain Intensity and Pain Related Disability (NRS-I)
Description: Study was terminated by VA. No VA outcome data to report.
Time Frame: baseline, 3, 6, 9, and 12 months
Population: No data were analyzed due to termination of the study.
Arm/Group | + Mobile | Standard-of-care
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Description: One patient in the mobile+ arm withdrew from participation.
Arm/Group | + Mobile | Standard-of-care
Serious Adverse Events (participants affected / at risk) | 0/34 | 0/35
Other Adverse Events (participants affected / at risk) | 0/34 | 0/35

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes